CLINICAL TRIAL: NCT00538733
Title: A Phase II Study of Thalidomide (THALOMID®), Clarithromycin (BIAXIN®), Lenalidomide(REVLIMID®), and Dexamethasone (DECADRON®) for Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: Phase II Study of Thalidomide, Clarithromycin, Lenalidomide, and Dexamethasone for Newly Diagnosed Multiple Myeloma
Acronym: T-BiRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707009285; RV-MM-PI-238
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: myeloma; newly diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Lenalidomide; Clarithromycin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-BiRD Therapy (Experimental): All patients were treated with the same regimen, starting with T-BIRD therapy (Cycles 1-4).
  After 4 cycles, Patients with disease progression will be taken off study. Patients who achieve maximum response will receive maintenance. Patients who achieve VGPR or PR will be given T-BiRD for 2 cycles (cycles 5-6). After 6 cycles of T-BiRD, Patients who achieve maximum response will receive maintenance; those with disease progression will be taken off study; all other patients will receive BIRD.
  Patients who progress on BiRD will reinitiate T-BiRD. If disease progression continues after 2 cycles, patients will be taken off study.
  Patients in CR/sCR or that achieve a plateau of disease for > 2 cycles on BiRD or T-BiRD therapy will receive maintenance.
  Interventions: Drug: thalomid; Drug: lenalidomide; Drug: clarithromycin; Drug: dexamethasone

INTERVENTIONS:
Drug: thalomid — Cycles 1-4
  • Thalidomide (50mg daily for days 1-7, thereafter 100mg daily for days 8-28 of the first 28 day cycle. Thalidomide will then be given at 100mg/daily for days 1-28 for each subsequent cycle)
Drug: lenalidomide — During T-BIRD Phase (Cycles 1-4, 5-6, and in the case of T-BIRD re-initiation)
  • Lenalidomide (25 mg daily days 1-21 of every 28 day cycle)
  During BiRD phase • 25mg daily days 1-21 of every 28 day cycle)
  During Maintenance Phase
  • 25 mg daily for days 1-21 out of a 28 day cycle
Drug: clarithromycin — During T-BiRD Phase • Clarithromycin (500mg twice daily for each 28 day cycle)
  During BiRD Phase:
  • Clarithromycin (500mg twice daily for each 28 day cycle)
Drug: dexamethasone — During T-BIRD Phase (Cycles 1-4, 5-6, and in the case of T-BIRD re-initiation)
  • Dexamethasone (40 mg daily on day 1, 8, 15 and 22 of each 28 day cycle)
  During BiRD Phase:
  • Dexamethasone (40 mg daily on day 1, 8, 15 and 22 of each 28 day cycle)
  During Maintenance Phase
  • Dexamethasone 20 mg weekly (days 1,8, 15, 22 out of a 28 day cycle)

SUMMARY:
Study Objectives

1. Evaluate the efficacy of the combination of thalidomide (Thalomid®), clarithromycin (Biaxin®), lenalidomide (Revlimid®), and dexamethasone (Decadron®) as an induction therapy for patients with newly diagnosed multiple myeloma (MM).
2. Evaluate the efficacy of the addition of thalidomide (Thalomid®) to BiRD combination therapy as a therapy to increase the complete response rate for patients with newly diagnosed multiple myeloma.
3. Evaluate the safety of the combination of clarithromycin, lenalidomide, dexamethasone, and thalidomide as a therapy for patients with newly diagnosed MM

DETAILED DESCRIPTION:
This phase II study is a treatment program for patients with newly diagnosed multiple myeloma. Up to 25 patients will be enrolled. Patients who sign consent and fulfill all eligibility criteria will be enrolled to receive the following treatment plan:

T-BiRD Therapy:

Cycles 1-4

* Thalidomide (50mg daily for days 1-7, thereafter 100mg daily for days 8-28 of the first 28 day cycle. Thalidomide will then be given at 100mg/daily for days 1-28 for each subsequent cycle)
* Clarithromycin (500mg twice daily for each 28 day cycle)
* Lenalidomide (25 mg daily days 1-21 of every 28 day cycle) and
* Dexamethasone (40 mg daily on day 1, 8, 15 and 22 of each 28 day cycle)
* Prophylactic medications will be given.

After completing 4 cycles

* Patients who demonstrate progression of disease will be taken off study.
* Patients who achieve maximum response (either by achievement of complete remission or stable disease plateau) will be transitioned to maintenance therapy.
* Patients who achieve VGPR or PR with acceptable toxicity will be given T-BiRD for an additional 2 cycles: cycles 5 and 6.

Upon completion of 6 cycles of T-BiRD,

* Patients who achieve maximum response (either by achievement of complete remission or stable disease plateau) will be transitioned to maintenance therapy.
* Patients without disease progression or maximum response (either by achievement of complete remission or stable disease plateau) will receive BiRD therapy
* Patients with disease progression will be taken off study.

BiRD therapy will consist of the following:

* Clarithromycin (500mg twice daily for each 28 day cycle)*
* Lenalidomide (25mg daily days 1-21 of every 28 day cycle)*
* Dexamethasone (40mg on days 1, 8, 15, 22 of each 28 day cycle)*
* Prophylactic medications will be continued.

  * Patients who finished T-BiRD therapy at reduced doses of clarithromycin, lenalidomide or dexamethasone will start BiRD therapy at the same doses of clarithromycin, lenalidomide and dexamethasone on which they ended T-BiRD therapy.

Patients who progress on BiRD will reinitiate T-BiRD as follows:

* Thalidomide (100mg/daily for days 1-28 for each 28 day cycle)
* Clarithromycin (500mg twice daily for each 28 day cycle)*
* Lenalidomide (25mg/daily for days 1-21 of each 28 day cycle)*
* Dexamethasone (40mg days 1, 8, 15, 22 of each 28 day cycle)*
* Prophylactic medications will be continued
* Patients who continue to show disease progression after two cycles of T-BiRD will be taken off study.

  * Patients who finished BiRD therapy at reduced doses of clarithromycin, lenalidomide or dexamethasone will start T-BiRD therapy at the same doses of clarithromycin, lenalidomide and dexamethasone on which they ended BiRD therapy.

Transition to maintenance therapy:

Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in quantitative M-spike as detected on serum immunofixation) for > 2 cycles on either BiRD or T-BiRD therapy will be transitioned to maintenance therapy. Maintenance therapy will be comprised of:

* Dexamethasone 20 mg weekly (days 1,8, 15, 22 out of a 28 day cycle)*
* Lenalidomide 25 mg daily for days 1-21 out of a 28 day cycle. (15mg daily will be given days 1 - 21 out of a 28 day cycle to patients with a creatinine clearance of < 40cc / minute).*
* Prophylactic medications will be continued

  * Patients who finished induction therapy with BiRD or T-BiRD at reduced doses lenalidomide or dexamethasone will start maintenance therapy at the same doses lenalidomide and dexamethasone on which they ended induction therapy. For patients with a creatinine clearance of < 40cc / minute, the lenalidomide dose will be the lower of their last induction therapy dose or 15mg daily on days 1 - 21 out of a 28 day cycle.

At the end of every cycle (which may coincide with day 1 of the new cycle), response and toxicity will be evaluated. During cycle 1, patients will have lab work done weekly (CBC with differential and blood electrolytes) and female of childbearing potential will have their pregnancy testing done, see APPENDIX III. All patients will remain on study until disease progression or side effects become excessive. Patients who achieve a stable plateau and are on maintenance therapy as defined above may be taken off study if eligible to proceed to high dose chemotherapy and autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Age > 18 years at the time of signing the consent form.
* Histologically confirmed Salmon-Durie stage II or III MM. Stage I MM patients will be eligible if they display poor prognostic factors (ß2M ≥5.5 mg/L, plasma cell proliferation index ≥5%, albumin of less then 3.0, and unfavorable cytogenetics).
* Newly diagnosed myeloma.
* No anti-myeloma therapy within 14 days prior to initiation of study treatment except for corticosteroids with a maximum allowed dosage equivalent to three pulses of dexamethasone (40mg daily for 4 days equals one pulse). Patients may be receiving adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care.
* Measurable disease as defined by > 1.0 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Karnofsky performance status ≥70% (>60% if due to bony involvement of myeloma.
* Able to take aspirin daily as prophylactic anticoagulation. (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* All study participants must be registered into the mandatory RevAssist® and S.T.E.P.S.® programs, and be willing and able to comply with the requirements of RevAssist® and the S.T.E.P.S.® programs.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide and thalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
* Life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥1000 cells/mm3 (1.0 x 109/L)
  * Platelets count ≥ 75,000/mm3 (75 x 109/L)
  * Serum SGOT/AST <3.0 x upper limits of normal (ULN)
  * Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  * Serum creatinine <2.5 mg/dL (221 µmol/L)
  * Serum total bilirubin <2.0 mg/dL (34 µmol/L)

Exclusion Criteria:

* Patients with non-secretory MM (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine).
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ≥ 5 years.
* Myocardial infarction within 6 months prior to enrollment , or NYHA(New York Hospital Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Pregnant or lactating females are ineligible.
* Given the potential of the study drugs to trigger or worsen HIV viremia and the incidence of opportunistic infections inpatients infected with the HIV virus, HIV-1 or HIV-2 positive patients will be excluded. The interactions of HAART with study drugs have not been determined.
* Active hepatitis B or hepatitis C infection.
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any coexisting medical problem or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial.
* Known hypersensitivity to dexamethasone, clarithromycin, lenalidomide, or thalidomide.
* History of thromboembolic event within the past 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Mark TM, Bowman IA, Rossi AC, Shah M, Rodriguez M, Quinn R, Pearse RN, Zafar F, Pekle K, Jayabalan D, Ely S, Coleman M, Chen-Kiang S, Niesvizky R. Thalidomide, clarithromycin, lenalidomide and dexamethasone therapy in newly diagnosed, symptomatic multiple myeloma. Leuk Lymphoma. 2014 Dec;55(12):2842-9. doi: 10.3109/10428194.2014.896005. Epub 2014 Mar 25. PMID 24576165

RESULTS

PARTICIPANT FLOW:
Groups:
- T-BiRD Therapy (All Patients): 26 patients started the treatment phase. Per protocol, completion of the treatment phase was defined as removal from treatment due to progression, or to pursue an alternative treatment (either a stem cell transplant, or further consolidation chemotherapy in pursuit of a transplant).
Period: Overall Study
Arm/Group | T-BiRD Therapy (All Patients)
Started | 26
Removed Due to Progression of Disease | 1
Removed to Pursue a Stem Cell Transplant | 11
Removed to Pursue Alternative Theray | 2
Completed | 14
Not Completed | 12
Not completed — Adverse Event | 8
Not completed — Death | 1
Not completed — declined to participate | 2
Not completed — still on therapy | 1

BASELINE CHARACTERISTICS:
Groups:
- T-BiRD Therapy (All Patients): All patients that enrolled on the study and received treatment with T-BiRD are included in this analysis.
Arm/Group | T-BiRD Therapy (All Patients)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 4
Durie-Salmon Classification [Number; unit: participants] — The Durie Salmon Staging System was used to assess patients clinical status. Stage 1A is associated with a better outcome and a low tumor burden, stage 2A is associated with a intermediate outcome and tumor burden, and stage 3A is associated with a worse outcome and higher tumor burden. Patients are classified into each stage based on multiple criteria including hemoglobin and calcium values, disease burden, and renal function.
  The Durie Salmon Staging System can be found here: https://www.themmrf.org/multiple-myeloma/prognosis/myeloma-stages/durie-salmon-staging-system/
  participants
    Stage 1A | 12
    Stage 2A | 9
    Stage 3A | 5
Cytogenetics [Number; unit: participants] — Cytogenetic analysis was done on all patients to determine if they were of standard or high risk. Cytogenetics were performed on bone marrow cultures.
  Standard risk was defined by the presence of one or more of the following on : t(11;14); hyperdiploidy; del 13q14 detected using florescence in situ hybridization (FISH); no abnormality High risk was defined by the presence of one or more of the following: del 17p; karyotype del 13q; amp 1q/del 1p; t(14;20); t(14;16); t(4;14)
  participants
    standard risk | 18
    high risk | 8
Immunoglobulins [Number; unit: participants]
  IgA myeloma | 3
  IgG myeloma | 15
  light chain only myeloma | 8
karnofsky performance status [Number; unit: participants] — Normal, no complaints = 100%; Able to carry on normal activities. Minor signs or symptoms of disease = 90%; Normal activity with effort = 80%; Care for self. Unable to carry on normal activity or to do active work = 70%; Requires occasional assistance, but able to care for most of his needs= 60% Requires considerable assistance & frequent medical care = 50%; Disabled. Requires special care & assistance = 40%; Severely disabled. Hospitalization indicated though death nonimminent = 30%; Very Sick, hospitalization necessary. Active supportive treatment necessary = 20%; moribund =10%; dead = 0%
  participants
    90% (or better) | 12
    80% | 12
    70% | 2
International Staging System Classification [Number; unit: participants] — Stage I ß2-M < 3.5 mg/dL and albumin =3.5 g/dL
  Stage II Neither stage I nor stage III
  Stage III ß2-M ≥ 5.5 mg/L
  participants
    Stage I | 9
    Stage II | 13
    Stage III | 4
Hemoglobin at baseline (in g/dL) [Median (Full Range); unit: g/dL] | 11.95 [9.1 to 15.4]
serum creatinine at baseline (in mg/dL) [Median (Full Range); unit: mg/dL] | 0.85 [0.5 to 1.9]
platelet count at baseline (in 1000/uL) [Median (Full Range); unit: 1000/uL] | 241 [87 to 383]
absolute neutrophil count at baseline (in 1000/uL) [Median (Full Range); unit: 1000/uL] | 3 [0.9 to 3.4]
albumin at baseline (in mg/dL) [Median (Full Range); unit: mg/dL] | 3.5 [2.2 to 4.4]
lactage dehydrogenase at baseline (U/L) [Median (Full Range); unit: U/L] | 151 [92 to 280]
C-reactive protein at baseline (in mg/dL) [Median (Full Range); unit: mg/dL] | 0.225 [0.03 to 10.3]
Beta-2 microglobulin at baseline (in mg/L) [Median (Full Range); unit: mg/L] | 2.2 [1.2 to 7.6]

OUTCOME MEASURES:

1. Primary Outcome: Effect of Drug Combination on Multiple Myeloma
Description: Objective response rate, defined according to the International Myeloma Working Group (IMWG) criteria as greater then or equal to a Partial Response (PR). The best response was recorded. The IMWG criteria can be found here: imwg.myeloma.org/international-myeloma-working-group-imwg-uniform-response-criteria-for-multiple-myeloma/
Time Frame: This was collected from patients for their duration on study treatment. Only the best response was recorded. Best responses were reported at any point of the study, from start of treatment up until removal of study, which occurred up to 57.4 cycles
Population: 25 of the 26 patients enrolled were accessible for response/progression, as one patient expired prior to first response assessment and could not be included in the analysis.
Measure: Number; unit: participants
Groups:
- T-BiRD Therapy (All Patients): 26 patients started the treatment phase. Per protocol, completion of the treatment phase was defined as removal from treatment due to progression, or to pursue an alternative treatment (either a stem cell transplant, or further consolidation chemotherapy in pursuit of a transplant). 25 of the 26 patients enrolled were accessible for response/progression, as one patient expired prior to first response assessment and could not be included in the analysis.
Arm/Group | T-BiRD Therapy (All Patients)
Number analyzed (Participants) | 25
participants
  sCR (stringent complete response) | 2
  VGPR (very good partial response) | 9
  PR (partial response) | 9
  SD (stable disease) | 5

2. Secondary Outcome: Median Time to Maximum Response
Description: Median Time to maximum response, reported in cycles of treatment. One cycle = 28 days.
Time Frame: from baseline to cycle with maximum response
Population: as for outcome 1
Measure: Median (Full Range); unit: cycles
Groups:
- T-BiRD Therapy (All Patients): 25 of the 26 patients enrolled onto the were assessed for response/progression, as one patient expired prior to first response assessment and could not be included in the analysis.
Arm/Group | T-BiRD Therapy (All Patients)
Number analyzed (Participants) | 25
cycles | 4 [1 to 7]

3. Secondary Outcome: Event Free Survival
Time Frame: from baseline to the time of first event that lead to removal from study (defined as progression, death, withdrawal of consent, or removal for toxicity)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- T-BiRD Therapy (All Patients): All 26 patients that were enrolled onto the study were assessed for event free survival.
Arm/Group | T-BiRD Therapy (All Patients)
Number analyzed (Participants) | 26
months | 21.5 [4.2 to 57.4]

4. Secondary Outcome: Progression Free Survival
Description: Progression determined using International Myeloma Working Group criteria, as defined below.
  An increase of > 25% from lowest response value one or more of the following:
  * Serum M-component and/or (the absolute increase must be > 0.5 g/dL)*
  * Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
  * Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL
  * Bone marrow plasma cell percentage; the absolute percentage must be > 10%
  * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder *if starting serum M protein is greater then 5 g/dL, absolute increase of 1g/dL is sufficient to determine relapse.
Time Frame: From start of treatment, to the date of first progression
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- T-BiRD Therapy (All Patients): 25 of the 26 patients enrolled onto the were assessed for progression, as one patient expired prior to first response assessment and could not be included in the analysis.
Arm/Group | T-BiRD Therapy (All Patients)
Number analyzed (Participants) | 25
months | 35.6 [14.1 to NA] — n/a has been entered because this was not reached

ADVERSE EVENTS:
Time Frame: Adverse events (serious and non-serious) were recorded from first dose of study drug, until removal from study (treatment).
Groups:
- T-BiRD Therapy (All Patients): All 26 patients that were enrolled onto the study were assessed for adverse events.
Arm/Group | T-BiRD Therapy (All Patients)
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-BiRD Therapy (All Patients) (N=26)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1
dizziness/fall (General disorders) | 1
atrial fibrillation (Blood and lymphatic system disorders) | 1
rash (steven johnson syndrome) (Skin and subcutaneous tissue disorders) | 1
multiple compression fractures (Musculoskeletal and connective tissue disorders) | 1
renal insufficiency/Congestive heart failure (Renal and urinary disorders) | 1
chest pain (Musculoskeletal and connective tissue disorders) | 1
deep vein thrombosis (Vascular disorders) | 1
myocardial infarction (Cardiac disorders) | 1
upper respiratory infection (Infections and infestations) | 1
sepsis (Infections and infestations) | 1
fever (Infections and infestations) | 1 — accompanied by dysgeusia and rash
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T-BiRD Therapy (All Patients) (N=26)
lymphopenia (Blood and lymphatic system disorders) | 26
neutropenia (Blood and lymphatic system disorders) | 8
anemia (Blood and lymphatic system disorders) | 6
thrombocytopenia (Blood and lymphatic system disorders) | 3
leukopenia (Blood and lymphatic system disorders) | 2
skin rash (Skin and subcutaneous tissue disorders) | 14
unspecified infection (Infections and infestations) | 11
anorexia/dysgeusia (Metabolism and nutrition disorders) | 10
dizziness (General disorders) | 7
hyperglycemia (Metabolism and nutrition disorders) | 5
psychomotor agitation (Psychiatric disorders) | 2
deep vein thrombosis (Vascular disorders) | 1
bacterial pneumonia (Infections and infestations) | 1
weakness (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less